CLINICAL TRIAL: NCT07136194
Title: Risk Factors of Postoperative Acute Kidney Injury and Mortality Among Hospitalized Patients Undergoing Major Surgery
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Li Yang, Professor, Peking University First Hospital
Other Study IDs: 2023-625-002
Record Dates: First submitted 2025-07-22; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Acute Kidney Injury; Major Surgery Under General Anesthesia; Mortality; Postoperative Complication; Risk Factors
Keywords: acute kidney injury; major surgery; mortality
MeSH Terms: conditions — Acute Kidney Injury; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients undergoing major surgery: Adult patients undergoing major surgery

SUMMARY:
The goal of this retrospective observational study is to learn about the intervenable risk factors of postoperative acute kidney injury (AKI) and in-hospital mortality among adult patients undergoing major surgery. The main questions it aims to answer are:

1. Does preoperative usage of potential nephrotoxic medications (eg., proton pump inhibitor, non-steroidal anti-inflammatory drugs) increase the risk of postoperative AKI and in-hospital mortality?
2. Does preoperative status (eg., malnutrition, hypoalbuminemia, hypomagnesemia) increase the risk of postoperative AKI and in-hospital mortality?
3. Are there intervenable risk factors of postoperative AKI and in-hospital mortality?
4. Are there special risk factors of postoperative AKI and in-hospital mortality in specific patients (eg. elderly, diabetics)? The study will be conducted in retrospective cohort of patients undergoing major surgery. Participants are followed until discharge.

DETAILED DESCRIPTION:
Acute Kidney Injury (AKI), characterized by a rapid decline of kidney function, is a common but serious postoperative complication in surgical patients, with an incidence ranging from 5.3% to 18.4%. Postoperative AKI is associated with increased mortality, prolonged hospital stays, and higher medical costs. Survivors are also prone to developing chronic kidney disease (CKD) or even end-stage renal disease (ESRD) . Identifying intervenable risk factors of postoperative AKI can help clinicians develop targeted strategies for high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* Hospitalized at Peking University First Hospital (PKUFH) between January 1, 2018, and December 31, 2020
* Undergoing major surgery during hospital stay

Exclusion Criteria:

* With fewer than two serum creatinine (SCr) measurements during hospitalization, or lack of postoperative SCr assessment
* With pre-exsiting CKD G5 (including long-term dialysis, prior/current kidney transplantation, or baseline estimated glomerular filtration rate [eGFR]<15mL/min/1.73m^2) at admission
* Undergoing radical or partial nephrectomy during current hospitalization
* Developing AKI prior to surgery or within 24 hours after admission (with admission diagnosis of AKI or meeting AKI criteria within 24 hours)
* With hospital stay < 24 hours

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive hospitalized adult patients (≥18 years) undergoing major surgery at Peking University First Hospital (PKUFH) between January 1, 2018, and December 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 21533 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative acute kidney injury | within 7 days after major surgery
  Acute kidney injury was defined by the KDIGO criteria. Postoperative AKI referred to acute kidney injury occurring within 7 days after major surgery.

SECONDARY OUTCOMES:
In-hospital acute kidney injury | after major surgery until up to 1year
  Acute kidney injury was defined by the KDIGO criteria. In-hospital acute kidney injury referred to acute kidney injury occurring after major surgery before discharge.
In-hospital mortality | after major surgery until up to 1 year
  death during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, Doctor, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The datasets are not publicly available as they are protected by Peking University First Hospital. Access requests should be directed to the principal investigator.